CLINICAL TRIAL: NCT01417026
Title: Promoting Social Perceptual Learning With Oxytocin in Autism
Brief Title: Intranasal Oxytocin and Learning in Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Schultz (Other)
Responsible Party: Sponsor-Investigator, Robert Schultz, Robert T. Schultz, PhD, Director of the Center for Autism Research, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-008241
Record Dates: First submitted 2011-08-11; First posted 2011-08-16 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism Spectrum Disorders; Oxytocin; Clinical Trial; Computer-based Intervention; Social Perception; Social Motivation; Social Cognition
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Oxytocin (Active Comparator): * Intranasal oxytocin (Trade name: Syntocinon)
  * Pharmacological class: The pharmacologic and clinical properties of Syntocinon are identical with the naturally occurring hormone oxytocin, which is released from the posterior pituitary.
  * Route of administration: Intranasal
  * Planned exposure: Each participant will receive one dose of intranasal oxytocin (24 IU) per day for 5 days.
  * One dose of 24 IU equals 6 spray puffs (3 puffs in each nostril).
  * Oxytocin will be imported from Victoria Pharmacy Zurich- Switzerland.
  Interventions: Drug: Intranasal Oxytocin (Trade name: Syntocinon)
- Intranasal Placebo (Placebo Comparator): * Intranasal placebo
  * The placebo is identical to the oxytocin formulation with the exception of the active compound.
  * Route of administration: Intranasal
  * Planned exposure: Each participant will receive one dose of intranasal placebo per day for 5 days.
  * One dose equals 6 spray puffs (3 puffs in each nostril).
  * Placebo will be imported from Victoria Pharmacy Zurich- Switzerland.
  Interventions: Drug: Intranasal Oxytocin (Trade name: Syntocinon)

INTERVENTIONS:
Drug: Intranasal Oxytocin (Trade name: Syntocinon) — This is a double-blind placebo-controlled trial of intranasal oxytocin in children and adolescents with ASD. Subjects will be randomized to 24 IU intranasal oxytocin or placebo for a 5 day period with concomitant game play of computer games, which are designed to enhance face perception skills. Measures of social function and cognition will be administered before and after the intervention period.
  Other Names: Syntocinon

SUMMARY:
The main objective of this study is to determine the safety and therapeutic potential of intranasal oxytocin in children and adolescents with autism spectrum disorder (ASD) when paired with a computer game intervention that is designed to enhance face perception skills.

DETAILED DESCRIPTION:
Recognizing faces is critical to social functioning, and can be improved for individuals with ASD by using intervention software in the form of appropriately designed computer games. The effects of this type of social intervention may be amplified with the concurrent use of oxytocin. Furthermore, these learning effects may impact social skills in general and translate to the level of the individual's everyday social behavior. Thus, the objective of this study is to determine the safety and therapeutic potential of intranasal oxytocin in children and adolescents with ASD when paired with a computer game intervention that is designed to enhance face perception skills.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 12-17 years, Mental age ≥ 10
2. Gender: males
3. Diagnosis of an Autism Spectrum Disorder
4. Consent: parent/guardian permission and child assent.
5. Ability to complete tasks: adequate vision, motor control of a keyboard and mouse, and fluency in English (and English as a first language).
6. Study participant needs to be clinically stable, in the opinion of the study clinicians. Stability will be assessed by the clinicians based on information from and conversations with the parent, if necessary. The parent needs to commit verbally to not making any changes to his or her child's current treatments for the duration of this study.

Exclusion Criteria:

1. History of traumatic brain injury, epilepsy/seizure disorder (except febrile seizures), or other significant medical, genetic, or neurological abnormality affecting growth, development, or motor or higher cortical functioning. Sensory impairments (e.g., significant vision/hearing loss).
2. Patients with one or more of the following: Human immunodeficiency virus (HIV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), hemophilia (bleeding problems, recent nose and brain injuries), abnormal blood pressure (hypotension or hypertension), drug abuse, immunity disorder, or severe depression.
3. Sensory impairments (e.g., significant vision/hearing loss).
4. Gestational age below 35 weeks and/or perinatal injury.
5. Profound mental retardation (e.g., Intelligence quotient (IQ) < 45) or sensory-motor difficulties that would preclude valid use of diagnostic instruments.
6. Lack of impairment in face recognition as determined by average or above average performance on the Benton Face Recognition Task.
7. Female participants.
8. Patients who are sensitive to Syntocinon or any components of its formulation.
9. Fever at the time of the baseline visit, defined as temperature above 37.5 degrees Celsius or 99.5 degrees Fahrenheit.
10. Judgment by the study physician or the PI that the patient is not suitable for the study due to unforeseeable safety issues.

Ages: 12 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2011-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert T. Schultz, PhD, Principal Investigator — Center for Autism Research, The Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of enrolled participants in the study was 36, but only 29 of those subjects were randomized. The 7 subjects who were not randomized did not meet study diagnostic or cognitive inclusion criteria.
Groups:
- Intranasal Oxytocin: * Intranasal oxytocin (Trade name: Syntocinon)
  * Pharmacological class: The pharmacologic and clinical properties of Syntocinon are identical with the naturally occurring hormone oxytocin, which is released from the posterior pituitary.
  * Route of administration: Intranasal
  * Planned exposure: Each participant will receive one dose of intranasal oxytocin (24 IU) per day for 5 days.
  * One dose of 24 IU equals 6 spray puffs (3 puffs in each nostril).
  * Oxytocin will be imported from Victoria Pharmacy Zurich- Switzerland.
  Intranasal Oxytocin (Trade name: Syntocinon): This is a double-blind placebo-controlled trial of intranasal oxytocin in children and adolescents with ASD. Subjects will be randomized to 24 IU intranasal oxytocin or placebo for a 5 day period with concomitant game play of computer games, which are designed to enhance face perception skills. Measures of social function and cognition will be administered before and after the intervention period.
- Intranasal Placebo: * Intranasal placebo
  * The placebo is identical to the oxytocin formulation with the exception of the active compound.
  * Route of administration: Intranasal
  * Planned exposure: Each participant will receive one dose of intranasal placebo per day for 5 days.
  * One dose equals 6 spray puffs (3 puffs in each nostril).
  * Placebo will be imported from Victoria Pharmacy Zurich- Switzerland.
  Intranasal Oxytocin (Trade name: Syntocinon): This is a double-blind placebo-controlled trial of intranasal oxytocin in children and adolescents with ASD. Subjects will be randomized to 24 IU intranasal oxytocin or placebo for a 5 day period with concomitant game play of computer games, which are designed to enhance face perception skills. Measures of social function and cognition will be administered before and after the intervention period.
Period: Overall Study
Arm/Group | Intranasal Oxytocin | Intranasal Placebo
Started | 16 | 13
Completed | 14 | 13
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Oxytocin | Intranasal Placebo | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 13 | 27
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 13 | 27
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Post-testing (After Max. 12 Days) on the Part/Whole Identity Test (LFI Skills Battery)
Description: This test measures the extent to which the participant employed a featural or holistic face recognition strategy. A sample face is presented, followed by a test face composed of either two whole faces or two face parts.
Time Frame: Baseline and Post-testing (after max. 12 days)
Measure: Mean (Standard Deviation); unit: change in percent correct
Arm/Group | Intranasal Oxytocin | Intranasal Placebo
Number analyzed (Participants) | 14 | 13
change in percent correct | 3.30 (10.78) | 3.17 (8.17)

2. Primary Outcome: Change From Baseline to Post-testing (After Max. 12 Days) on the Reading the Mind in the Eyes Test (Child Version)
Description: This is a test of emotion recognition. This test asks children to pick the best word out of four options to describe the mental state of a set of eyes. The test includes 28 photographs of eyes with both affective (e.g., upset) and cognitive (e.g., thoughtful) mental state words as choices.
Time Frame: Baseline and Post-testing (after max. 12 days)
Measure: Mean (Standard Deviation); unit: change in items correct
Arm/Group | Intranasal Oxytocin | Intranasal Placebo
Number analyzed (Participants) | 12 | 11
change in items correct | 0.33 (3.92) | 1.82 (3.34)

3. Secondary Outcome: Changes From Baseline to Post-testing (After Max. 12 Days) on the "Happy Faces" Measure of Social Attention
Description: The "Happy Faces" task requires that participants look at a series of faces of men and women. Faces are presented on the screen one by one and children are asked just to look at the faces. Eye movements are measured with a Tobii x120 tabletop eye-tracker to evaluate participants' looking patterns towards the eyes versus the mouth region.
Time Frame: Baseline and Post-testing (after max. 12 days)
Measure: Mean (Standard Deviation); unit: change in proportion of looking
Arm/Group | Intranasal Oxytocin | Intranasal Placebo
Number analyzed (Participants) | 8 | 9
change in proportion of looking
  looking to faces relative to full screen | .02 (.18) | -0.05 (.25)
  looking to objects relative to full screen | -.03 (.14) | .08 (.18)

ADVERSE EVENTS:
Time Frame: 12 Days
Arm/Group | Intranasal Oxytocin | Intranasal Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 11/16 | 12/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intranasal Oxytocin (N=16) | Intranasal Placebo (N=13)
Cold-like symptoms (i.e. runny nose, stuffy nose, sneezing) (General disorders) | 6 | 3
Burning and irritation of sinuses (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bloody nose (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased sense of smell (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Ear aches/hot ears (Ear and labyrinth disorders) | 0 | 2
Breathing problems (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eyes (burning, watery, teary, aching, etc.) (Eye disorders) | 3 | 2
Headaches (Nervous system disorders) | 0 | 4
Rapid pounding heart (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Diarrhea, soft bowels, sore stomach (Gastrointestinal disorders) | 1 | 1
Tongue ulcer and gum pain (Gastrointestinal disorders) | 0 | 1
Flaking scalp (Skin and subcutaneous tissue disorders) | 1 | 0
Frustration, cranky, agitation (Psychiatric disorders) | 4 | 3
Tired, Exhausted, Fatigued, decreased energy level, felt sedated (Psychiatric disorders) | 4 | 1
Increased energy level, hyperactivity (Psychiatric disorders) | 1 | 1
Nervous feeling (Psychiatric disorders) | 1 | 1
Increased awareness and social interaction (Psychiatric disorders) | 1 | 1
Increased appetite (Psychiatric disorders) | 1 | 0
Hand wringing (Psychiatric disorders) | 0 | 1
Sleep problems (Psychiatric disorders) | 0 | 1
Strange physical feelings (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes